CLINICAL TRIAL: NCT01213654
Title: Pain Relief After VATS Lobectomy Using Interoperatively Placed Inter Costal Catheters.
Brief Title: Inter Costal Catheters for Video-Assisted Thoroscopic (VATS) Lobectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Dept. of thoracic Surgery (Ambiguous); Dept. of cardio-thoracic anaesthesia (Ambiguous); Dept. Surgical PAthophysiology (Ambiguous); all Blegdamsvej 9, 2100-Copenhagen, Denmark (Unknown)
Responsible Party: MD Kim Wildgaard, Section for Surgical Pathophysiology
Other Study IDs: VATS-IC-2010
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Lung Cancer Patients
Keywords: Lung cancer; VATS Lobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A pilot study to observe satisfaction of analgesia with intercostal catheters after VATS lobectomy.

DETAILED DESCRIPTION:
Pain and satisfaction with pain treatment is investigated in a population after VATS lobectomy.

ELIGIBILITY:
Inclusion Criteria:

Age of consent (ie age>=18) Eligible for lobectomy Able to comply Willing to register postoperatively

-

Exclusion Criteria:

* do not understand DAnish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting lung cancer patients due for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
NRS (pain score 0-10)) | Until discharge (2-4 days)
  Painscore
satisfaction (Verbal ranking scale 1-4) | until discharge, 2-4 days
  qualitative measurement

SECONDARY OUTCOMES:
Side effects (quantitatively, see details) | until discharge, 2-4 days
  Daily presence of, Nausea Dizziness Vomiting Sedation Pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark